CLINICAL TRIAL: NCT01090193
Title: Phase 4 Study :Human Kidney Histopathology in Acute Obstructive Jaundice: a Prospective Study
Brief Title: Human Kidney Histopathology in Obstructive Jaundice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turkish Ministry of Health Izmir Teaching Hospital (Other Government)
Responsible Party: Assoc. Prof. Adam Uslu/ Chief of the Department of General Surgery, Turkish Ministry of Health Izmir Teaching Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BZYK01
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2009-01

CONDITIONS: Patients With Obstructive Jaundice
Keywords: Obstructive jaundice; kidney histopathology; lactulose
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- obstructive jaundice (Other)
  Interventions: Procedure: Whipple operation,Hepaticojejunostomy

INTERVENTIONS:
Procedure: Whipple operation,Hepaticojejunostomy — Whipple operation, Hepaticojejunostomy
  Other Names: Internal biliary drainage operations

SUMMARY:
Introduction: Cholemia and bacterial translocation with portal endotoxemia are integral in the pathogenesis of obstructive jaundice (OJ). There is sufficient experimental data about hemodynamic and histopathologic consequences of OJ. On the contrary, pathologic information of renal changes in patients with OJ is still lacking. Therefore; the primary objective of this prospective study is to demonstrate the specific histopathologic changes in kidneys of patients with short-term biliary tract obstruction receiving a standard perioperative medical treatment protocol.

DETAILED DESCRIPTION:
Twenty consecutive patients with biliary obstruction were included. Fluid replacement, prevention of biliary sepsis and portal endotoxemia were mainstays of the perioperative treatment protocol. Fluid and electrolyte balance was maintained by twice daily body weight calculations, central venous pressure and mean arterial pressure (MAP) monitoring . Renal function was assessed by glomerular filtration rate estimation via MDRD-7 formula.

Kidney biopsy evaluation was focused on tubular changes, thrombotic microangiopathy, endothelial damage and peritubular capillary (PTC) dilatation with or without C4d staining. Fresh frozen sections were evaluated with immunoflourescence (IF)microscopy for glomerular IgG, IgA, IgM, C3, and C1q staining.

Despite those favourable figures, dilatation of peritubular venules and acute tubular necrosis were demonstrated synchronously in all cases. C4d staining in PTC and arterioles and thrombotic microangiopathy were entirely absent in the study group. Immune complex deposits in peritubular capillaries and in glomeruli were not detected. Three patients had isolated glomerular C4d deposition without accompanying thrombotic microangiopathy and IgG, IgA, IgM, C3, and C1q staining of glomerular capillaries in IF microscopy.

Discussion: This study is the first in the literature to address the histopathologic changes that occur in humans with short-term biliary obstruction. ATN and venous dilatation was observed in all biopsies, without exception, despite the maintenance of strict volume control in all patients. The adequacy of volume control may not be implicated in those results; rather a possible mechanism related to untrapped endotoxin in the gut lumen or systemic circulation might lead to prolonged peritubular capillary dilatation and hypoperfusion with synchronous acute tubular necrosis . Absolute recovery of renal function in all patients and the demonstration of solitary ATN with no microvascular-glomerular-interstitial inflammation or injury, suggests that the perioperative treatment regime in this study is fairly efficacious in short-term OJ.

ELIGIBILITY:
Inclusion Criteria:

* Between January 2009 and January 2010, twenty consecutive patients with an equal distribution of biliary obstruction type (10 malignant and 10 benign) were included into the study.

Exclusion Criteria:

* Patients over 60 years of age or those with a history of co-morbid cardiac disease were initially evaluated by echocardiography.
* Those with an ejection fraction rate <50% and left ventricular end-diastolic diameter (LVDD) over 52 mm. were excluded from the study because of the already existing left ventricular dysfunction compromising the optimisation of fluid replacement.
* Patients with a history and serologic evidence of acute/chronic parenchymal kidney or liver disease were also excluded.

Ages: 26 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Human kidney histopathology in acute obstructive jaundice: a prospective study | 12 months
  the primary objective of this prospective study is to demonstrate the specific histopathologic changes in kidney parenchyme of patients undergoing surgery for short-term biliary tract obstruction.

SECONDARY OUTCOMES:
Human kidney histopathology in acute obstructive jaundice: a prospective study | 12 months
  The secondary objective is to approve the feasibility of a standard perioperative medical treatment protocol, which has been implemented on a routine basis in our department over the last decade.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Uslu, Assoc. Prof., Principal Investigator — Izmir Teaching Hospital
Locations (1):
- Izmir Teaching Hospital, Department of General Surgery, Izmir, Turkey (Türkiye)

REFERENCES:
- [Result] Green J, Better OS. Systemic hypotension and renal failure in obstructive jaundice-mechanistic and therapeutic aspects. J Am Soc Nephrol. 1995 May;5(11):1853-71. doi: 10.1681/ASN.V5111853. PMID 7620083